CLINICAL TRIAL: NCT00000684
Title: Continuous High-Dose Intravenous Dextran Sulfate in Human Immunodeficiency Virus-Infected Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 105; 11080 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Infusions, Intravenous; Dextran Sulfate; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Dextran Sulfate

INTERVENTIONS:
Drug: Dextran sulfate

SUMMARY:
To determine the safety and effectiveness of dextran sulfate when it is administered intravenously at the maximum tolerated dose (MTD) as a treatment for HIV infection in AIDS patients. The effect of dextran sulfate on platelet survival will also be assessed in 3 patients to help determine the mechanism of thrombocytopenia (low platelets) noted in all patients receiving intravenous dextran sulfate in this study.

Dextran sulfate appears to inhibit HIV in experiments in the test tube, but studies conducted in humans to determine its effect on HIV when dextran sulfate is given orally have not been conclusive. It is hoped that this study will show that dextran sulfate administered intravenously

DETAILED DESCRIPTION:
Dextran sulfate appears to inhibit HIV in experiments in the test tube, but studies conducted in humans to determine its effect on HIV when dextran sulfate is given orally have not been conclusive. It is hoped that this study will show that dextran sulfate administered intravenously will have antiviral effects in patients who are infected with HIV.

Following tests for evaluation, patients are hospitalized for 14 days. They are admitted to the hospital in the afternoon and, starting the next morning, receive a continuous infusion of dextran sulfate through an intravenous line for 14 days. The infusion is adjusted to maintain an activated partial thromboplastin time (APTT) of 50 to 65 seconds. Blood is withdrawn 5 times on the first day that patients receive dextran sulfate and at least once a day thereafter for safety. Patients' clinical condition, blood clotting, and blood platelets are monitored very closely.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acetaminophen.

Patients must have:

-

Clinically documented AIDS or AIDS-related complex (ARC) defined as CDC group IVA or history of any of the findings that define CDC group IV subgroup C-2:

* oral candidiasis, oral hairy leukoplakia, multidermatomal herpes zoster, recurrent nontyphoidal Salmonella bacteremia, or nocardiosis.

Prior Medication:

Allowed:

* Acetaminophen.

Exclusion Criteria

Concurrent Treatment:

Excluded:

* Intramuscular injections.

Patients will be excluded from the study for the following reasons:

* Acute illness requiring hospitalization or antiviral drug therapy for treatment.
* Volunteers who have taken any antiviral medications, anticoagulants, antiplatelet medications, or any nonsteroidal anti-inflammatory drugs, except acetaminophen, within 2 weeks of study entry, or those who anticipate the need for such medication during the study.
* Positive stool guaiac at screening.
* Disorders of coagulation or any known contraindication to anticoagulation, including but not limited to gastrointestinal or other serious bleeding, major trauma or surgery within the past 2 months, stroke or suspicion of central nervous system (CNS) bleeding, Kaposi sarcoma (with or without proven gastrointestinal involvement), and any known CNS lesions that might be prone to bleed.
* Allergy to dextran sulfate or heparin.
* Acute or asymptomatic HIV infection.

Prior Medication:

Excluded:

* Antiviral medications.
* Anticoagulants.
* Antiplatelet medications.
* Any nonsteroidal anti-inflammatory drugs (except acetaminophen).

Prior Treatment:

Excluded:

* Hospitalization for acute illness.

Patients may not have any of the following diseases or symptoms:

* Allergy to dextran sulfate or heparin.
* Acute or asymptomatic HIV infection.
* Acute illness requiring hospitalization.
* Chronic anemia requiring transfusion within the past month.
* Disorders of coagulation or any known contraindication to anticoagulation, including but not limited to gastrointestinal or other serious bleeding, major trauma or surgery within the past 2 months, stroke or suspicion of central nervous system (CNS) bleeding, Kaposi's sarcoma, and any known CNS lesions which might be prone to bleed.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Study Completion 1991-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lietman PS, Study Chair; Flexner CW, Study Chair
Locations (1):
- Johns Hopkins Adult AIDS CRS, Baltimore, Maryland, United States

REFERENCES:
- [Background] Flexner C, Barditch-Crovo PA, Kornhauser DM, Farzadegan H, Nerhood LJ, Chaisson RE, Bell KM, Lorentsen KJ, Hendrix CW, Petty BG, et al. Pharmacokinetics, toxicity, and activity of intravenous dextran sulfate in human immunodeficiency virus infection. Antimicrob Agents Chemother. 1991 Dec;35(12):2544-50. doi: 10.1128/AAC.35.12.2544. PMID 1810188